CLINICAL TRIAL: NCT03822624
Title: Randomized, Double Blind, Placebo Controlled Study to Evaluate Efficiency and Safety on the Use of a Probiotic in SCORAD Reduction in 4-to-17 Years-old Patients With Atopic Dermatitis
Brief Title: Study to Evaluate the Use of a Probiotic in SCORAD Reduction in Young Patients With Atopic Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biopolis S.L. (Industry)
Collaborators: Korott, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATOP/PRO-2
Record Dates: First submitted 2018-12-04; First posted 2019-01-30 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Atopic Dermatitis
Keywords: Probiotic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental)
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic mixture with three bacterial strains with maltodextrin as a carrier.
  Arms: Probiotic group
Other: Placebo — Placebo comparator with maltodextrin as a carrier.
  Arms: Placebo group

SUMMARY:
The study's objective is to confirm that an oral probiotic treatment reduces the signs and symptoms of moderate atopic dermatitis determined by SCORAD, in patients aged 4 to 17 years, as compared to placebo. It will also be examined if the probiotic treatment, as compared to placebo, reduces the quantity of topical steroids used to treat disease flares, and increases the time till the first disease flare after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 to 17 years, both inclusive.
* Diagnosed with atopic dermatitis according to Hanifin and Rajka criteria.
* SCORAD index of 20-40, both inclusive.
* Patients whose parents or legal guardian sign the informed consent.
* The minor over 12 years must also give their consent to participate in the trial.

Exclusion Criteria:

* Pregnancy.
* Breast feeding.
* Women of childbearing age who, in the opinion of the investigator, do not commit to using an effective method of contraception, if they have an active sex life or start during the trial.
* Treated with phototherapy for the atopic dermatitis in the previous 2 months.
* Treated with systemic corticosteroids in the previous 2 months or need for corticosteroids anticipated during the first 12 weeks of the study.
* Having undergone cytotoxic or immunosuppressive therapy in the previous 2 months or having an anticipated need for cytotoxic or immunosuppressive therapy during the first 12 weeks of the study.
* Treated with probiotics in the previous two months.
* Treated with systemic antibiotics in the previous four days.
* Patients with a fever (temperature > 37.5°C, axillary or equivalent).
* Serious allergic diseases.
* Diseases related to immunodeficiency processes or cancer.
* Other skin diseases that can make assessment of the atopic dermatitis difficult or which require the continuous use of topical corticosteroids.
* Patients in whom any of the study products is contraindicated according to its summary of product characteristics.
* Patients who have participated in research studies with medicinal products during the previous 3 months.
* Patients with gluten or lactose intolerance or inflammatory bowel disease (Crohn's disease or ulcerative colitis).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the SCORAD index at 12 weeks. | 12-week
  SCORAD: SCOring of Atopic Dermatitis
  Subscales:
  Eczema Spread (A): 0 - 20 Eczema Intensity (B): 0 - 63 Subjective Symptoms (C): 0 - 20
  Total = (A/5) + (Bx7/2) + C Total: 0 - 103 (Higher values represent a worse outcome)

SECONDARY OUTCOMES:
Number of days that each patient requires the administration of topical corticosteroids. | 12-week
Number of days that each patient requires the administration of topical corticosteroids in disease flares. | 12-week
Total dose of topical corticosteroids. | 12-week
Number of patients who reach a CGI score lower than 2. | 12-week
  CGI: Clinical Global Impression
  Total: 0 - 5 (Higher values represent a worse outcome)
Number of adverse events. | 12-week
Use of antihistamines and other treatments. | 12-week
Adherence to the treatment. | 12-week
  Percentage of treatment intake days.
Disease-free time up to 24 weeks. | 24-week

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Quirónsalud San José, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Vithas Nisa 9 de Octubre, Valencia